CLINICAL TRIAL: NCT00362843
Title: PET Measurement of Regional Rates of Cerebral Protein Synthesis in Subjects With Fragile X Syndrome
Brief Title: Protein Synthesis in the Brain of Patients With Fragile X Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060214; 06-M-0214
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Fragile X Syndrome; Healthy Volunteers
Keywords: 11C-Leucine; Positron Emission Tomography (PET); Cerebral Protein Synthesis; dexmedetomidine; Brain Mapping; Natural History; Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: healthy volunteers
- patients: Patients with Fragile X Syndrome
  Interventions: Drug: [15-O]water

INTERVENTIONS:
Drug: [15-O]water
  Groups: patients

SUMMARY:
Biosynthesis of proteins is essential for growth and continued maintenance of the entire neuron including axons, dendrites, and synaptic terminals, and it is clearly one of the important biochemical processes underlying adaptive changes in the nervous system. Studies in experimental animals with the quantitative autoradiographic L [1 (14)C]leucine method have demonstrated a number of the physiological and pathological conditions in which changes in regional rates of cerebral protein synthesis (rCPS) occur.

We have recently developed the first fully quantitative method for determining rCPS with positron emission tomography (PET). The PET method was adapted from the autoradiographic L [1 (14)C]leucine method; it uses L [1 (11)C]leucine as the PET tracer, dynamic scanning, and a kinetic modeling approach for quantification. This method was validated in nonhuman primates by comparison of PET measurements with those based on established biochemical and autoradiographic techniques.

The objective of the present study is to examine the degree to which changes in rCPS in human subjects can be quantified with the L [1 (11)C]leucine PET method. We propose three studies to be carried out sequentially. In Part I we will establish the L-[1-(11)C]leucine PET method in human subjects. In Part II we will measure rCPS in normal control subjects in two states: awake and under deep sedation/general anesthesia with propofol. A difference in rCPS between these two states may indicate that we can detect activity-dependent protein synthesis with the PET method. In Part III we will study subjects with fragile X syndrome. This patient group was chosen since the affected gene in fragile X syndrome codes for a protein that is thought to be a negative regulator of message translation. Thus an effect on protein synthesis may be very close to the underlying genetic abnormality in fragile X syndrome. Regionally selective increases in rCPS have been found in studies in a mouse model of this disease.

The present study will establish the sensitivity of the L [1 (11)C]leucine PET method to detect changes in rCPS in human subjects. A quantitative and sensitive method to measure rCPS with PET will augment the tools available for investigating the brain and its regional adaptive responses. Ultimately the method may have widespread applications, not only for the study of normal development and plasticity but also in clinical medicine, e.g., in the investigation of disorders of brain development, recovery from brain injury, and neurodegenerative diseases.

SPECIFIC AIMS

1. <TAB>Establish the L-[1-(11)C]leucine PET method for measurement of rCPS in human subjects. Evaluate the optimal scan time and the variability of the measurement in an individual.
2. <TAB>Determine the effect of deep sedation with propofol on rCPS in normal human subjects. We will use the [1-(11)C]leucine PET method to evaluate lambda, i.e., the fraction of the precursor pool for protein synthesis that is derived from arterial plasma, and rCPS in the same subjects under awake and deep sedation conditions.

   I)<TAB>Hypothesis 1a. Deep sedation with propofol has effects on rCPS.

   II)<TAB>Hypothesis 1b. Deep sedation with propofol has effects on values of lambda.
3. <TAB>Assess the sensitivity of the [1-(11)C]leucine PET method to detect differences in rCPS in subjects with fragile X syndrome.

I)<TAB>Hypothesis 3a. There are regionally selective changes in rCPS in subjects with fragile X syndrome compared with age-matched healthy controls. Regions affected include hippocampus, thalamus, hypothalamus, amygdala, and frontal and parietal cortex.

II)<TAB>Hypothesis 3b. In centrum semiovale, cerebellum, striatum and occipital and temporal cortex rCPS are unchanged in subjects with fragile X syndrome compared with age-matched healthy controls.

III)<TAB>Hypothesis 3c. Values of lambda in the brain as a whole and in the regions examined are unchanged in subjects with fragile X syndrome compared with age-matched healthy controls.

IV) Hypothesis 3d. The average rate of protein synthesis in the brain as a whole is unchanged in subjects with fragile X syndrome compared with age-matched healthy controls.

DETAILED DESCRIPTION:
Biosynthesis of proteins is essential for growth and continued maintenance of the entire neuron including axons, dendrites, and synaptic terminals, and it is clearly one of the important biochemical processes underlying adaptive changes in the nervous system. Studies in experimental animals with the quantitative autoradiographic L-[1-(14)C]leucine method have demonstrated a number of the physiological and pathological conditions in which changes in regional rates of cerebral protein synthesis (rCPS) occur.

We have recently developed the first fully quantitative method for determining rCPS with positron emission tomography (PET). The PET method was adapted from the autoradiographic L-[1-(14)C]leucine method; it uses L-[1-(11)C]leucine as the PET tracer, dynamic scanning, and a kinetic modeling approach for quantification. This method was validated in nonhuman primates by comparison of PET measurements with those based on established biochemical and autoradiographic techniques.

The objective of the present study is to examine the degree to which changes in rCPS in human subjects can be quantified with the L-[1-(11)C]leucine PET method. Three studies will be carried out sequentially. In Part I we have established the L-[1-11C]leucine PET method in human subjects. Three studies to be carried out sequentially. In Part I we will establish the L-[1-(11)C]leucine PET method in human subjects. In Part II we measured rCPS in normal control subjects in two states: awake and under deep sedation/general anesthesia. A difference in rCPS between these two states may indicate that we can detect activity-dependent protein synthesis with the PET method. In Part III we will study subjects with fragile X syndrome. This patient group was chosen since the affected gene in fragile X syndrome codes for a protein that is thought to be a negative regulator of message translation. Thus an effect on protein synthesis may be very close to the underlying genetic abnormality in fragile X syndrome. Regionally selective increases in rCPS have been found in studies in a mouse model of this disease.

The present study establishes the sensitivity of the L-[1-(11)C]leucine PET method to detect changes in rCPS in human subjects. A quantitative and sensitive method to measure rCPS with PET will augment the tools available for investigating the brain and its regional adaptive responses. Ultimately the method may have widespread applications, not only for the study of normal development and plasticity but also in clinical medicine, e.g., in the investigation of disorders of brain development, recovery from brain injury, and neurodegenerative diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Fragile X subjects:

Male subjects, 18-24 years of age, with diagnosis of fragile X syndrome will be considered. Diagnosis will be confirmed by molecular genetic testing. Subjects with CGG repeat sequences greater than 200 and methylation of FMR1 will be included.

Control:

Male subjects, 18-24 years of age will be considered.

EXCLUSION CRITERIA:

Fragile X subjects:

Fragile X subjects with a high level of repeat size or methylation mosaicism will be excluded. Fragile X subjects on psychotropic medications will be excluded from the study. Fragile X subjects who have received radiation doses for research purposes exceeding 4 rem (whole body effective dose) in the previous 12 months will be excluded. Fragile X subjects in whom MRI is contraindicated will be excluded. Subjects with metal objects in their bodies, such as pacemakers, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses, cochlear implants, or shrapnel fragments will be excluded from the study. Welders and metal workers at risk for eye injury because of unsuspected tiny metal fragments there will also be excluded. Subjects in whom sedation is contraindicated will be excluded. Fragile X subjects on medications that interfere with blood coagulation will be excluded (see Appendix 1). In addition, fragile X subjects with respiratory illnesses or cardiovascular diseases will be excluded as there might be increased risk of complications with sedation/anesthesia.

Control:

Subjects with premutation alleles, i.e., repeat length between 55 and 200 will be excluded. Subjects with IQ less than 90 or subnormal language skills will be excluded. Subjects on psychotropic medication will be excluded from the study. Subjects who have received radiation doses for research purposes exceeding 3.5 rem (whole body effective dose) in the previous 12 months and subjects for whom MRI is contraindicated will be excluded. Subjects in whom sedation is contraindicated will be excluded from Part II. Subjects on medications that interfere with blood coagulation will be excluded (see Appendix 1). Subjects with any previous history of psychiatric or neurological disease, as assessed by the Structured Clinical Interview for DSM-IV (SCID), will be excluded. In addition, subjects with respiratory illnesses or cardiovascular diseases will be excluded from Part II as there might be increased risk of complications with sedation/anesthesia. Subjects positive for HIV will be excluded from the study. Subjects with positive results on the urine drug screen will be excluded.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: All of our subjects are adult, male volunteers between the ages of 18 and 24, either healthy volunteers or patients with Fragile X Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2006-08-22 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Regional rates of cerebral protein synthesis | ongoing
  regional rates of cerebral protein synthesis

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen L, Toth M. Fragile X mice develop sensory hyperreactivity to auditory stimuli. Neuroscience. 2001;103(4):1043-50. doi: 10.1016/s0306-4522(01)00036-7. PMID 11301211
- [Background] Coenen HH, Kling P, Stocklin G. Cerebral metabolism of L-[2-18F]fluorotyrosine, a new PET tracer of protein synthesis. J Nucl Med. 1989 Aug;30(8):1367-72. PMID 2787848
- [Background] Davis HP, Squire LR. Protein synthesis and memory: a review. Psychol Bull. 1984 Nov;96(3):518-59. No abstract available. PMID 6096908
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-M-0214.html